CLINICAL TRIAL: NCT05987527
Title: Long-Term Follow-Up of Patients Who Have Received an Autologous Antigen-Specific Chimeric Antigen Receptor T Regulatory Cell Therapy (CAR- Treg Therapy, TX200-TR101) in a Prior Clinical Study
Brief Title: Long-Term Follow-Up of TX200-TR101 (STEADFAST Long Term)
Status: Active, not recruiting | Type: Observational
Sponsor: Sangamo Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: TX200-KT03; 2022-002440-40 (EudraCT Number)
Record Dates: First submitted 2023-06-30; First posted 2023-08-14 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Kidney Transplant Rejection; End Stage Renal Disease
Keywords: Regulatory T-Cells; Genetically modified cells; Chimeric antigen receptor; Long term follow up; T-Regs; Cell Therapy
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment group: Subjects underwent a kidney transplant as per planned standard of care and were administered study drug TX200-TR101 in study TX200-KT02 post transplantation
  Assigned interventions - subjects who received TX200-TR101 in clinical study TX200-KT02
  Interventions: Diagnostic Test: Blood sample
- Control group: Subjects underwent a kidney transplant as per planned standard of care in study TX200-KT02 with no study drug administered
  Interventions: Diagnostic Test: Blood sample

INTERVENTIONS:
Diagnostic Test: Blood sample — Routine procedures

SUMMARY:
This long-term follow-up study is being conducted to collect long-term (up to 15 years post-infusion) safety and tolerability data from subjects enrolled in studies evaluating TX200-TR101.

DETAILED DESCRIPTION:
This is long- term follow up observational trial for patients who participated previously to a multicentre, first-in-human, open-label, single ascending dose, dose-ranging study of autologous, chimeric antigen receptor T regulatory cells (CAR-Treg) in HLA-A2 mismatched living donor kidney transplant recipients, with a control cohort of mismatched kidney transplant recipients of similar immunological risk.

The aim is for this observational long-term follow up study (TX200-KT03) is to collect long-term (up to 15 years post-infusion) safety and tolerability data from subjects enrolled in studies evaluating TX200-TR101.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who enrolled in the Phase I/IIa study TX200-KT02, received a transplanted kidney and have either completed or withdrawn from that study.
2. Willing and able to provide written informed consent (IC) in accordance with local regulations and governing Independent Ethics Committee (IEC)/Institutional Review Board (IRB) requirements prior to any procedure or evaluation performed specifically for the sole purpose of the study.

Exclusion Criteria:

* N/A

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Transplant recipients enrolled in the Phase I/IIa study (TX200-KT02) and who have consented to participate in this LTFU study,
Sampling Method: Non-Probability Sample
Enrollment: 11 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2039-06-11 (Estimated); Study Completion 2039-06-11 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of TX200-TR101 infusion evaluated by overall survival | Up to 15 years post infusion
  Long term safety and tolerability of TX200-TR101 infusion evaluated by overall survival
Safety and Tolerability TX200-TR101 infusion evaluated by and incidence of serious adverse events (SAEs) according to CTCAE V5.0. | Up to 15 years post infusion
  Long term safety and tolerability of TX200-TR101 infusion evaluated by and incidence of serious adverse events (SAEs) according to CTCAE V5.0.

SECONDARY OUTCOMES:
Long term graft related outcomes | Up to 15 years post infusion
  Incidence of graft rejection according to the Banff classification criteria
Number of in-patient days in hospital to evaluate the effect of TX200-TR101 over a long term | Up to 15 years post infusion
  Number of in-patient days in hospital
Incidence of Adverse Events related to TX200-TR101 over a long term period | Up to 15 years post infusion
  Incidence of Adverse Events related to TX200-TR101
Incidence of Adverse Events of special interest as defined in the protocol over long term | Up to 15 years post infusion
  Incidence of Adverse Events of special interest as defined in the protocol
Change in immunosuppression regime to evaluate long term safety of TX200-TR101 | Up to 15 years post infusion
  Change in immunosuppression regime
Incidence of graft loss due to rejection to evaluate the composite efficacy profile of TX200-TR101 | Up to 15 years post infusion
  Incidence of graft loss due to rejection
Incidents of deaths to evaluate composite efficacy profile of TX200-TR101 | Up to 15 years post infusion
  Incidences of death of TX200-TR101 participants
Incidence of chronic graft dysfunction measured by changes in estimated glomerular filtration rate to evaluate the composite efficacy profile of TX200-TR101 | Up to 15 years post infusion
  Incidence of chronic graft dysfunction measured by changes in estimated glomerular filtration rate

CONTACTS AND LOCATIONS:
Locations (5):
- University Hospitals Leuven, Leuven, Belgium
- Netherlands (3):
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Centre, Leiden
  - Erasmus MC, University Medical Center, Rotterdam
- Oxford University Hospitals NHS Foundation Trust, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to parent study STEADFAST, TX200-KT02 — https://clinicaltrials.gov/ct2/show/NCT04817774?term=TX200-KT02&draw=2&rank=1